CLINICAL TRIAL: NCT07141758
Title: Investigation of Salivary E-cadherin, Calprotectin, and Matrix Metalloproteinase-9 Levels in Patients With Recurrent Aphthous Stomatitis
Brief Title: Salivary E-cadherin, Calprotectin, and Matrix Metalloproteinase-9 Levels in Recurrent Aphthous Stomatitis
Status: Recruiting | Type: Observational
Sponsor: Selin Yeşiltepe (Other)
Collaborators: Aydın Adnan Menderes University Scientific Research Projects Unit (Unknown); Aydin Adnan Menderes University (Other)
Responsible Party: Sponsor-Investigator, Selin Yeşiltepe, Associate Professor, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Other Study IDs: 2025/02
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Aphthous Stomatitis; Aphthous Ulcer
Keywords: E-cadherin; Calprotectin; MMP-9; ELISA; Recurrent aphthous stomatitis; RAS; Saliva; Salivary Biomarkers
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Unstimulated whole saliva samples will be collected using Salivette® saliva collection swabs (Sarstedt, Germany) from all participants. After centrifugation, the supernatant (clear fluid portion) will be separated and transferred into sterile Eppendorf tubes. These saliva supernatant samples will be stored at -80°C and retained for the analysis of proteins (E-cadherin, Calprotectin, and MMP-9) using ELISA. No DNA will be extracted or used from the samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minor Recurrent Aphthous Stomatitis Patients: Participants aged 18 years or older who have been clinically diagnosed with minor recurrent aphthous stomatitis (RAS) based on characteristic clinical features and medical history. The lesion must be round or oval, less than 5 mm in diameter, surrounded by an erythematous halo, and covered by a grayish-white pseudomembrane. Eligible patients must have experienced at least three episodes of RAS within the past year and present with at least one aphthous ulcer at the time of clinical examination and saliva collection.
  Interventions: Diagnostic Test: ELISA
- Healthy Controls: Participants aged 18 years or older with no lifetime history of recurrent aphthous stomatitis. Control group participants will be selected to match the patient group in terms of age and gender distribution. At the time of saliva collection, no aphthous lesions or any active oral mucosal pathology should be present.
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — Unstimulated saliva samples will be non-invasively collected from participants in this study to measure the concentrations of E-cadherin, Calprotectin, and MMP-9. These protein concentrations will be quantified using commercially available Enzyme-Linked Immunosorbent Assay (ELISA) kits.

SUMMARY:
The goal of this observational cross-sectional study is to determine the salivary levels of E-cadherin, Calprotectin, and Matrix Metalloproteinase-9 (MMP-9) in patients with Recurrent Aphthous Stomatitis (RAS) and to compare them with those of healthy controls.

The main questions it aims to answer are:

Are the salivary levels of E-cadherin, Calprotectin, and MMP-9 significantly different in patients with minor RAS compared to healthy controls?

Can these salivary proteins serve as biomarkers involved in the pathogenesis of minor RAS?

Researchers will compare patients with minor RAS and healthy individuals to determine whether differences in salivary E-cadherin, Calprotectin, and MMP-9 levels are associated with the presence of disease.

Participants will:

Provide unstimulated saliva samples using a saliva swab

Undergo clinical evaluation for periodontal status (Community Periodontal Index - CPI) and caries experience (DMFT index)

Collected saliva samples will be stored at -80°C until analysis. The concentrations of the investigated proteins will be measured using ELISA kits, and total protein levels will be determined using a colorimetric protein assay.

The relationships among the salivary concentrations of the investigated proteins, as well as their associations with demographic variables such as age and sex, will be analyzed.

DETAILED DESCRIPTION:
Hypotheses H₀ (Null Hypothesis): There is no statistically significant difference in salivary levels of E-cadherin, Calprotectin, and Matrix Metalloproteinase-9 (MMP-9) between patients with Recurrent Aphthous Stomatitis (RAS) and healthy controls.

H₁ (Alternative Hypothesis): There is a statistically significant difference in salivary levels of E-cadherin, Calprotectin, and MMP-9 between patients with RAS and healthy controls.

Sample Size Calculation Based on an effect size of 0.50, a power of 80%, and a type I error rate (α) of 5%, the required sample size for the study was calculated to be 102 participants using the "t tests - Means: Difference between two independent means (two groups)" module in G*Power (version 3.1).

Formation of Participant Groups Two study groups will be established: a patient group and a healthy control group. Patients clinically diagnosed with minor recurrent aphthous stomatitis (RAS) based on characteristic clinical appearance and medical history will be included in the patient group. For the diagnosis of minor RAS, a history of at least three episodes of RAS within the past year will be considered a required criterion. This lesion should be round or oval in shape, less than 5 mm in diameter, surrounded by an erythematous halo at the periphery, and covered by a grayish-white pseudomembrane. In order to obtain a salivary sample, at least one aphthous lesion must be present at the time of examination. Control group participants with a similar age and gender distribution and no lifetime history of RAS will be selected and included in the study.

In this study, the threshold value of DMFT < 5.0, defined by the World Health Organization (WHO) as a very low caries risk level in adults, will be used as an inclusion criterion for all participants.

DMFT Index:

D (Decayed): Number of decayed teeth M (Missing): Number of teeth lost due to caries F (Filled): Number of filled teeth due to past caries T (Teeth): Total number of teeth evaluated Participants with DMFT ≥ 5.0 will be excluded from the study. To assess periodontal status, the Community Periodontal Index (CPI) will be used. The CPI is a standardized system developed by the World Health Organization (WHO) to evaluate periodontal health. The index teeth (11, 16, 17, 26, 27, 31, 36, 37, 46, 47) will be examined to allow for rapid and standardized assessment of periodontal conditions. Periodontal measurements will be performed using the WHO Community Periodontal Index probe. Each index tooth will be assessed at four sites: buccal, lingual/palatal, mesial, and distal. The highest score recorded for each tooth or quadrant will be noted. The highest score in any quadrant will be used to represent the participant's overall CPI score.

0 - Healthy periodontal tissues

1. - Bleeding observed upon probing
2. - Calculus detected during probing
3. - Pocket depth of 4-5 mm
4. - Pocket depth of 6 mm or more If one of the two molars in the posterior quadrant is missing, it will not be replaced by another tooth. In cases where no suitable index teeth are available in a quadrant, all present teeth in that quadrant will be examined, and the highest score will be recorded as the quadrant's CPI score. The distal surfaces of third molars will not be included in the assessment. Only participants with a CPI score of 0-2 will be included in the study.

Collection and Analysis of Saliva Samples For saliva collection, the swab method, which is one of the unstimulated saliva collection techniques, will be used. Salivette® swab (Sarstedt, Germany) will be utilized to collect saliva samples from participants. In accordance with the manufacturer's instructions, samples will be taken at least 60 minutes after any food or drink intake (liquid or solid) or tooth brushing. Participants will be asked to rinse their mouths with water for 1-5 seconds approximately 10 minutes before sampling. They will then be instructed to hold the absorbent swab in their mouth without chewing for at least 2 minutes. After that, the swab will be removed and placed into the inner suspended tube of the Salivette container by the participant. Samples will be centrifuged within 4 hours using the A-PRF12 centrifuge (Germany) at 1000 × g for 2 minutes. During centrifugation, heavy particles (cells, debris, or other precipitable materials) will settle at the bottom of the tube, while the lighter, soluble components will remain in the upper phase (supernatant). Following centrifugation, the supernatant portion of the saliva will be carefully separated and transferred to sterile Eppendorf tubes. The samples will be coded and stored at -80°C until biochemical analysis. After all samples have been collected, they will be transferred to the Department of Biochemistry, Faculty of Medicine, Aydın Adnan Menderes University, and analyzed using the ELISA method on the same day. Human E-cadherin, Human MMP-9, and Human CALP (Calprotectin) ELISA kits, along with the BCA Protein Colorimetric Assay Kit, will be used according to the manufacturer's instructions. The concentrations of the investigated proteins as well as total protein levels will be measured in the saliva samples. The concentration of each investigated protein will be normalized by calculating its ratio to the total salivary protein concentration. This normalization will account for inter-sample variability due to differences in salivary flow rate, cellular content, or sample volume.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older
* Clinically diagnosed with minor recurrent aphthous stomatitis (RAS) (defined as having a history of at least three RAS episodes within the past year)
* Systemically healthy (i.e., without any diagnosed systemic disease)
* No history of tobacco use
* Presence of at least one active aphthous ulcer at the time of saliva sample collection
* No known mental or physical disabilities

Exclusion Criteria:

* Use of any pharmacological treatment within the past 3 months
* Use of antiseptic mouthwash within the past 3 months
* Pregnant or lactating individuals, or those currently using oral contraceptives
* History of systemic diseases associated with oral ulcerations such as Crohn's disease, ulcerative colitis, celiac disease, or Behçet's disease
* History of chemotherapy or radiotherapy
* Current or prior use of immunomodulatory drugs, cytotoxic agents, or systemic corticosteroids
* Undergoing orthodontic treatment (to avoid misdiagnosis with traumatic ulcers)
* Use of removable dental prostheses (to avoid misdiagnosis with traumatic ulcers)
* Presence of periodontal disease (CPI score of 3 or 4)
* Caries risk not classified as very low (DMFT ≥ 5)
* Presence of pathological oral mucosal lesions such as lichen planus, pemphigus vulgaris, or mucous membrane pemphigoid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a total of 102 participants, including 51 patients clinically diagnosed with minor recurrent aphthous stomatitis (RAS) and 51 healthy controls. All participants will be aged 18 years or older. Patients must have experienced at least three episodes of minor RAS within the past year and present with at least one active aphthous ulcer at the time of saliva collection. Only systemically healthy, non-smoking individuals without periodontal disease or oral mucosal pathology will be included. Control group participants will be matched by age and gender to the patient group and must have no lifetime history of RAS.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Salivary Concentrations of E-cadherin, Calprotectin, and Matrix Metalloproteinase-9 (MMP-9) Using ELISA | Baseline (single visit)
  The concentrations of E-cadherin, Calprotectin, and MMP-9 in unstimulated saliva samples will be measured using the Enzyme-Linked Immunosorbent Assay (ELISA) technique. Commercially available human ELISA kits will be used in accordance with the manufacturers' instructions. The analysis will be performed on the saliva supernatant collected from each participant, and results will be reported in ng/mL. Saliva samples will be collected from two groups:
  Minor Recurrent Aphthous Stomatitis (RAS) patients: Patients who present with at least one active aphthous ulcer at the time of saliva collection.
  Healthy controls: Participants without current aphthous lesions or any other active oral mucosal pathology at the time of saliva collection.

SECONDARY OUTCOMES:
Total Salivary Protein Concentration Using Bicinchoninic Acid (BCA) Colorimetric Assay | Baseline (single visit)
  Total protein concentration in unstimulated saliva samples will be measured using the Bicinchoninic Acid (BCA) Protein Colorimetric Assay Kit, following the manufacturer's protocol. The resulting values (expressed in mg/mL) will be used both for quantification and for normalizing the concentrations of investigated proteins (E-cadherin, Calprotectin, and MMP-9). This measure will help control for variability in salivary flow rate, sample volume, or protein content across participants. Minor Recurrent Aphthous Stomatitis (RAS) patients: Patients who present with at least one active aphthous ulcer at the time of saliva collection. Healthy controls: Participants without current aphthous lesions or any other active oral mucosal pathology at the time of saliva collection.

CONTACTS AND LOCATIONS:
Overall Officials: Selin Yeşiltepe, dds,msd, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koray M, Atalay B, Akgul S, Oguz FS, Mumcu G, Saruhanoglu A. Relationship between salivary calprotectin levels and recurrent aphthous stomatitis: A preliminary study. Niger J Clin Pract. 2018 Mar;21(3):271-275. doi: 10.4103/njcp.njcp_23_17. PMID 29519972